CLINICAL TRIAL: NCT04346238
Title: Characterization of the Interruptions of the GAA Expansion and Study of Their Influence on the Severity of Friedreich's Ataxia : INTREP-AF
Brief Title: Characterization of the Interruptions of the GAA Expansion and Study of Their Influence on the Severity of Friedreich's Ataxia
Acronym: INTREP-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Neurogenetic department, CHU Bordeaux (Unknown); Genetic Department , CHU Montpellier-France (Unknown); Neurology department, CHU La réunion (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0029
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Friedreich Ataxia
Keywords: Neurology; Genetic; Friedreich ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Friedriech Ataxia genetically confirmed: Patients with Friedriech Ataxia genetically confirmed
  Interventions: Other: Reuse of existing data from patients' medical records

INTERVENTIONS:
Other: Reuse of existing data from patients' medical records — Reuse of existing data from patients' medical records

SUMMARY:
Friedreich's ataxia (FA) is the most frequent recessive genetic ataxia with an estimated prevalence of 1/50 000. The first symptoms appear around the age of 10 years with a progressive course and the need for an armchair 10- 15 years after the first symptoms. More rarely the disease can present with a late onset (after the age of 25) with a picture characterized by spastic paraparesis and slower progression ("LOFA" for "Late Onset Friedreich Ataxia" or VLOFA for "Very Late Appearance of Friedreich's ataxia ").

AF is caused in 96% of cases by an expansion of GAAN triplets (N> 100 repeats) located in intron 1 of the FXN gene, present on the two alleles, and, in the rest of the cases, by an associated expansion a point mutation or a deletion in trans. During molecular diagnostics, it is not uncommon to find the presence of interruptions within the GAA expansion. This results in the absence and / or the shift of peak (s) within the chromatogram.

To date, only the partial correlation between the size of the expansion and the age of onset of Friedreich's ataxia has been established. In particular, very atypical forms of AF with a late onset (after the age of 25) are in particular explained by the low number of repetitions in the expansion, typically between 100 and 500 repetitions. However, the presence of an interruption could stabilize the size of the expansion and, therefore, be mainly associated with expansions of small sizes and therefore with a late onset of the disease.

The objective of this study is therefore to analyse and caracterize the presence and the type of interruptions of the GAA expansions in a group of patients with FA ; this data will be correlated with the age at onset of FA.

ELIGIBILITY:
Inclusion criteria:

* Subjects with diagnosis of genetically confirmed Friedreich's Ataxia (AF) and :
* two expansions of GAAN triplets (> 100 repetitions or "premutation", corresponding to> 32 but <100 repetitions) located in intron 1 of the FXN gene present on the two alleles;
* symptomatic (SARA scale> 4);
* having signed a consent for the performance of genetic analyzes which also includes the authorization for the conduct of further studies for research purposes and the authorization for the collection, entry and computer processing of medical data, in all confidentiality. A newsletter on the principle of non-opposition will be sent.

Exclusion criteria:

* Patients with Friedreich's ataxia due to an expansion associated with a point mutation or a deletion in trans;
* Patients who, at the time of signing the genetic consent, objected to the use of their data for research purposes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Friedriech Ataxia genetically confirmed. .
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Interruptions and date at onset | 18 months
  Study the correlation between the presence and type of interruptions (location within the expansion, nucleotide sequence: "GAAA", "GAG", etc.) and the age of onset of Friedreich's ataxia.

SECONDARY OUTCOMES:
Clinical correlation | 18 months
  Estimate the interaction between the presence and type of interruption and the age of onset of the various functional impacts (walking, cardiac involvement).

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Marelli, MD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC